CLINICAL TRIAL: NCT00693914
Title: Working Memory Performance Among Childhood Brain Tumor Survivors Treated With Conformal Radiation Therapy: A Pilot Study
Brief Title: Working Memory Performance Among Childhood Brain Tumor Survivors
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: EXFXN1; R21CA131616 (NIH)
Record Dates: First submitted 2008-06-05; First posted 2008-06-09 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2011-10

CONDITIONS: Brain Tumors
Keywords: Brain Tumor; Cognitive Late Effects; Radiation Therapy; Working Memory
MeSH Terms: conditions — Brain Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Brain Tumor Survivors (n=50)
  Interventions: Behavioral: Series of tests/questionnaires
- 2: Healthy Sibling Controls (n=40)
  Interventions: Behavioral: Series of tests/questionnaires
- Solid Tumor Survivors (n=40)
  Interventions: Behavioral: Series of tests/questionnaires

INTERVENTIONS:
Behavioral: Series of tests/questionnaires — Developmental and Demographic, KINDL Health-Related Quality of Life, Adaptive Behavior Assessment System (ABAS-II),Behavior Rating Inventory of Executive Function (BRIEF), Wechsler Digit Span Task, Wide Range Achievement Test 3rd Edition (WRAT3),Wechsler Abbreviated Scale of Intelligence (WASI), Pediatric Immediate Post-Concussion Assessment and Cognitive Testing (ImPACT), Recognition Memory Task: Face Stimuli, Recognition Memory Task: Verbal Stimuli, Self Ordered Search: Object, Self Order Search: Verbal

SUMMARY:
Children treated with radiation therapy for brain tumors are at risk for cognitive problems. These problems have typically been demonstrated on global cognitive measures including measures of intellectual functioning (IQ). Identification of specific areas of impairment can assist in isolating vulnerable brain areas and developing targeted interventions.

In this study, we assess brain tumor survivors, solid tumor controls and healthy sibling controls using measures of working memory (online maintenance and manipulation of information) in order to identify a specific cognitive process that may underlie the observed decline in IQ. We are also exploring relationships among working memory performance with IQ, clinical characteristics and a specific genetic factor of interest.

DETAILED DESCRIPTION:
This is a cross-sectional controlled study of brain tumor survivors treated at St. Jude with conformal radiation therapy. Brain tumor survivors (n= 50, solid tumor survivors (n=40), and healthy sibling controls (n= 40) are evaluated once only with laboratory measures of cognitive skills (working memory, episodic memory and estimated IQ) and parental questionnaires (executive and adaptive functions). We also use buccal (cheek) swabs to gather samples for DNA extraction. We hypothesize: brain tumor survivors will perform significantly worse than solid tumor and healthy controls on measures of working memory, working memory will correlate significantly with IQ, working memory will be associated with parent report of executive functions and a specified genotype related to dopamine metabolism will be associated with working memory impairment.

ELIGIBILITY:
Inclusion Criteria:

Brain Tumor Patients

* Treated for a primary central nervous system (CNS) tumor with conformal radiation therapy and enrolled on the institutional protocol RT-1
* Initiated radiation therapy at least 2 years prior to enrollment with no evidence of recurrent disease
* Age 8-18 years inclusive at the time of enrollment, with sampling to obtain a broad cross-section of participants in terms of age, tumor location and time since RT initiation
* English as the primary language
* Research participant and one parent willing to participate and provide consent/assent according to institutional guidelines

Solid Tumor Patient Controls

* Treated for a solid tumor (i.e., Ewing's sarcoma, osteosarcoma, soft tissue/rhabdomyosarcoma, neuroblastoma or Wilms tumor) at St. Jude without CNS directed therapy - Diagnosed at least 2 years prior to enrollment
* Age 8-18 inclusive at the time of enrollment, with age, gender and race sampling to broadly match the brain tumor group
* English as the primary language
* Research participant and one parent willing to participate and provide consent/assent according to institutional guidelines

Sibling Controls

* Healthy sibling controls- siblings of St. Jude patients treated for a brain tumor (not necessarily on RT-1)
* Age 8-18 inclusive, with age and gender sampling to broadly match the patient group
* English as a primary language
* Research participant and one parent willing to participate and provide consent/assent according to institutional guidelines

Exclusion Criteria:

Brain Tumor Patients

* Significant impairment in global intellectual functioning (operationalized as an estimated IQ less than 70 as indicated by most recent RT-1 testing)
* History of documented CNS injury or disease predating cancer diagnosis
* History of documented Attention Deficit Hyperactivity Disorder (ADHD) predating cancer diagnosis by at least one year (must have been diagnosed by a physician with medication prescribed)
* Treatment with psychostimulant or psychotropic medication within two weeks of study enrollment
* Sensory or motor impairment that would preclude valid cognitive testing

Solid Tumor and Sibling Controls

* Significant impairment in global intellectual functioning (operationalized as a history of special education in a self-contained classroom)
* History of documented CNS injury or disease
* History of documented Attention Deficit Hyperactivity Disorder (ADHD) (must have been diagnosed by a physician with medication prescribed)
* Treatment with psychostimulant or psychotropic medication within two weeks of study enrollment
* Sensory or motor impairment that would preclude valid cognitive testing

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Both the patient group and sibling group will be accrued using a broad stratification process for gender (Male, Female) and age (8-12 years of age, 13-18 years of age).
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2007-04; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Performance on experimental working memory measures (computerized self-ordered pointing tasks) | Collected during one time cross-sectional assessment.

SECONDARY OUTCOMES:
Abbreviated IQ (WASI), episodic memory measures (computerized word and face recognition tasks) and parent questionnaires of executive (BRIEF) and adaptive (ABAS-II) functioning. | Collected during one time cross-sectional assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Heather M Conklin, Ph.D., Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org